CLINICAL TRIAL: NCT06772077
Title: Safety and Usability of the ATLAS 2030 Exoskeleton in Pediatric Patients With Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other); Fundación del Lesionado Medular (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS-LM
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: Spinal Cord Injury; Rehabilitation; robotics; Gait Exoskeleton; children; ATLAS2030
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robot Asissted Gait Training (Experimental): The rehabilitation sessions will be carried out by a physiotherapist trained in rehabilitation with the ATLAS 2030 exoskeleton
  Interventions: Device: Rehabilitation treatment with ATLAS2030

INTERVENTIONS:
Device: Rehabilitation treatment with ATLAS2030 — 10 sessions of Rehabilitation Treatment with ATLAS2030 with With an evaluation session before the first session and another one after 10 sessions.
  Other Names: Robot Asissted Gait rehabilitation

SUMMARY:
The goal of this clinical trial is to analyze the usability and safety of the robotic gait ATLAS 2030 in a cohort of pediatric patients with Spinal Cord Injury, with the aim of extending its indication for use to pediatric spinal cord injury

DETAILED DESCRIPTION:
Spinal cord injury has a relatively low prevalence in the pediatric population, although its effects have significant physical and psychological consequences that greatly impact the quality of life of affected children. The ATLAS 2030 exoskeleton is a robotic gait device approved by the Spanish Agency of Medicines and Medical Devices for the rehabilitation of pediatric patients with cerebral palsy and spinal muscular atrophy. The principal aim is to analyze the safety and usability of the ATLAS 2030 exoskeleton during the implementation of a robotic gait training program with this device in a cohort of pediatric patients with spinal cord injury. the secondary aim is to analyze, in the same cohort of pediatric patients with spinal cord injury and through the implementation of the same therapeutic program, the efficacy of the ATLAS 2030 exoskeleton in improving fatigability, mood, health perception, and gait speed.

Ten sessions with the ATLAS 2030 exoskeleton will be conducted with pediatric patients with acute or chronic spinal cord injury. Additionally, two assessment sessions will be performed before and after the series of sessions.

ELIGIBILITY:
Inclusion Criteria:

* Having a subacute or chronic spinal cord injury (SCI) and being clinically stable with a general condition good enough to participate in the therapeutic program with the ATLAS 2030.
* Age between 3 and 14 years.
* Medical authorization to perform standing and gait training with weight-bearing.
* Consent from the participant or legal guardian to participate in the study.
* Adequate level of acceptance and commitment from the family.

Inclusion criteria related to device characteristics:

* Weight ≤ 35 kg.
* Hip width ≤ 34 cm. It is advised that for measurements under 28 cm, verification should be performed to ensure there is no excessive base of support that might induce foot inversion in the standing position.
* Femur length (distance from the greater trochanter to the lateral condyle of the femur) between 24 cm and 33 cm. Femur lengths shorter than 24 cm are acceptable as long as the hip motor of the device does not extend above the user's iliac crest, avoiding hypermobility of the lumbar spine.
* Tibia length (distance from the lateral condyle to the lateral malleolus of the tibia) between 23 cm and 32 cm. Tibia lengths shorter than 23 cm are acceptable as long as they can be compensated with a lift and the user's ankle joint remains within the area of the ankle motor.
* EU shoe size between 27 and 33.

Exclusion Criteria:

* Impossibility for the family to complete treatment schedule planning.
* Any contraindication for standing and/or walking.
* Spasticity (Modified Ashworth Scale (MAS) = 4 in the lower limbs at the time of device use).
* Joint contracture of the hip and/or knee > 20 degrees.
* Need to walk with more than 9 degrees of hip abduction.
* Need to walk with more than 9 degrees of dorsal or plantar ankle flexion, or inability to use an orthosis to achieve 90° at the ankle.
* Severe skin lesions in areas of contact with the device.
* Planned surgical intervention during the study period or previous orthopedic surgery on the spine and/or lower limbs contraindicating treatment.
* Known advanced osteoporosis evidenced by bone densitometry, particularly with a history of prior fractures or fractures without trauma. Traumatic bone fractures in the lower limbs or pelvic girdle within the past 6 months.
* Unstable fractures, joint dislocations, or other joint pathologies in the trunk and lower limbs contraindicating the treatment.
* Severe rigid orthopedic deformities of the spine that prevent the use of the device.
* Presence of frequent seizures, uncontrolled epilepsy, or difficult-to-control behavioral disorders.
* Presence of decompensated heart or lung disease, or any other condition causing exercise intolerance.
* Allergy to any of the materials used in the ATLAS 2030: cotton, nylon, polyester, polyamide, polyethylene, or polypropylene.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | From enrollment to the last assessment session at 8 weeks
  occurrence of any serious adverse event to the participant
Falls prevalence | From enrollment to the last assessment session at 8 weeks
  Number of falling events occurred from the participant or caregiver
Skin integrity | From enrollment to the last assessment session at 8 weeks
  Occurrence of any injury of the skin in the areas of contact and produced by the use of the device
Pain assessment | From enrollment to the last assessment session at 8 weeks
  pain measured by the Visual Analogic Scale (VAS) by the participant, scored from 0 to 10, being 0 "no pain" and 10 "unbearable pain"
Heart rate | from the beginning to the end of treatment at 6 weeks
  measurement of heart rate
Oxygen saturation | from the beginning to the end of treatment at 6 weeks
  measurement of Oxygen saturation when medical prescription
Blood pressure | from the beginning to the end of treatment at 6 weeks
  measurement of blood pressure. Systolic and diastolic pressures will be assessed
User and/or caregiver perception of the device | From enrollment to the last assessment session at 8 weeks
  Questions that are scored from 0 to 5 on aspects related to comfort, weight, volume, etc
Device usage data | From enrollment to the last assessment session at 8 weeks
  Total walking time. Unit of Measure: Minutes.
Number of steps | From enrollment to the last assessment session at 8 weeks
  Number of steps with the device
Usage modes | From enrollment to the last assessment session at 8 weeks
  two different usage modes (active and automatic).
Speed | From enrollment to the last assessment session at 8 weeks
  speed achieved with the device (steps per minute)
Range of motion | From enrollment to the last assessment session at 8 weeks
  Passive Degree to which a joint can move (hip, knee, and ankle joints in both legs). From 0º to 180º.

SECONDARY OUTCOMES:
State of mind | from the beginning to the end of treatment at 6 weeks
  It will be done with a Likert-type scale from 1 to 5 (1: very sad; 2: sad; 3: indifferent; 4: happy; 5: very happy). This scale will be administered before and after each therapeutic session.
Health perception | from enrollment to the last assessment session at 8 weeks
  EQ-5D scale assesses five dimensions of health: Mobility, Self-care, Usual activities, Pain/Discomfort, and Anxiety/Depression.
  Each dimension has five levels of severity (No problems, Slight problems, Moderate problems, Severe problems, and Extreme problems).
Health perception | from enrollment to the last assessment session at 8 weeks
  Visual Analogue Scale (VAS) is a vertical scale where patients rate their current health on a scale from 0 to 100 (0 representing "the worst health you can imagine" and 100 representing "the best health you can imagine.
10 Meter Walking Test (10 MWT) measured with ATLAS 2030 | From enrollment to the last assessment session at 8 weeks
  The 10 Meter Walking Test (10MWT) records the time taken by the participant to walk 10 meters with the device in motion intent mode.
Effort perception | from the beginning to the end of treatment at 6 weeks
  Borg Rating of Perceived Exertion (RPE), is a tool used to measure the intensity of physical activity based on how hard you feel your body is working.
  - Modified Borg Scale (0-10): This version ranges from 0 to 10, where 0 means "nothing at all" and 10 means "very, very hard." It's often used in clinical settings to assess symptoms like breathlessness, chest pain, and muscle fatigue.

OTHER OUTCOMES:
Classification of Spinal Cord Injury | From enrollment to the last assessment session at 8 weeks
  The International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) is a standardized tool for assessing and classifying spinal cord injuries Sensory function: Assessed in 28 dermatomes per side for light touch and pinprick sensations, scored as 0 (absent), 1 (impaired), or 2 (normal). Maximum score: 224 points (112 per modality).
  Motor function: Evaluated in 10 key muscle groups per side, using a 0-5 strength scale. Maximum score: 100 points.
  ASIA Impairment Scale: Classifies the severity of spinal cord injury into five categories: from A (complete) to E (normal).
Disability | From enrollment to the last assessment session at 8 weeks
  The Spinal Cord Independence Measure (SCIM) III. It is composed of 19 items that assess three main domains:
  * Self-care (6 items, scores range from 0-20)
  * Respiration and sphincter management (4 items, scores range from 0-40)
  * Mobility (9 items, scores range from 0-40) The total SCIM scores range from 0 to 100
Walking ability | From enrollment to the last assessment session at 8 weeks
  WISCI II (Walking Index for Spinal Cord Injury): Assess walking ability and level of assistance needed.
  Scoring: 0: Cannot walk. 20: Independent walking. Intermediate (1-19): Varies with assistive devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nacional Parapléjicos, Toledo, Spain